CLINICAL TRIAL: NCT05336487
Title: Physical Activity, Sports, and Health in Adults With Intellectual Disabilities
Brief Title: Physical Activity, Sports and Health in Adults With Intellectual Disabilities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Novo Nordisk A/S (Industry); Elsass Foundation (Other)
Responsible Party: Principal Investigator, Jacob Wienecke, Principal Investigator, Associate Professor, University of Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2553227/4242
Record Dates: First submitted 2022-03-31; First posted 2022-04-20 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Intellectual Disability
Keywords: Intellectual disability; Physical activity; Cardiovascular fitness; Bone health; Body composition
MeSH Terms: conditions — Intellectual Disability; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A physically active intervention group is compared to a physically inactive control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity group (PA-group) (Experimental): The intervention group. Participants with intellectual disabilities is recruited from a local daily activity center, where the participants participate in teacher-organized physical activity ~2 hours/day, 5 days/week.
  Interventions: Other: Physical activity
- Control Group (CON-group) (No Intervention): The control group. The participants with intellectual disabilities is recruited from daily activity centers, which does not use physical activity in their daily work with the participants.

INTERVENTIONS:
Other: Physical activity — 2 hours of physical activity per day, 5 days per week, for the intervention period
  Arms: Physical Activity group (PA-group)

SUMMARY:
Currently, there is a paucity of quality research within the field of health science with a focus on persons with intellectual disabilities, and especially how longer lasting periods of varied physical activity affects the target group. There is a lack of insight, in how persons with intellectual disabilities learns and retains movement skills. Thus, the research group behind this project will investigate the following research questions:

1. Does 40 weeks of intense and varied sports and physical activities as an intervention lead to positive changes in health status for adults with intellectual disabilities?
2. Can lasting effects be measured three and six months after the intervention?
3. Does the intervention improve the motor competences for the participants?
4. How does defined groups of adult persons with Down syndrome and Cerebral Palsy learn and retain a new motor skill?

ELIGIBILITY:
Inclusion Criteria:

* Presence of an intellectual disability

Exclusion Criteria:

* Participants under guardianship
* Unable to give informed consent to participate on their own

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in body weight | Measurements will be obtained at pre-intervention, (0 weeks), mid intervention (14 weeks) and post intervention (40 weeks)
  Body weight in kilograms
Change in body fat mass | Measurements will be obtained at pre-intervention, (0 weeks), mid intervention (14 weeks) and post intervention (40 weeks)
  Body fat mass in kilograms
Change in lean mass | Measurements will be obtained at pre-intervention, (0 weeks), mid intervention (14 weeks) and post intervention (40 weeks)
  Lean body mass in kilograms
Change in fat free mass | Measurements will be obtained at pre-intervention, (0 weeks), mid intervention (14 weeks) and post intervention (40 weeks)
  Fat free mass in kilograms
Change in cardiovascular fitness | Measurements will be obtained at pre-intervention, (0 weeks), mid intervention (14 weeks) and post intervention (40 weeks)
  Change in heart rate during the same absolute submaximal exercise intensity
Change in areal bone mineral density of the whole body | Measurements will be obtained at pre-intervention, (0 weeks), mid intervention (14 weeks) and post intervention (40 weeks)
  Areal bone mineral density in grams per square centimeter (g/cm2) of the whole body
Change in T-scores of the whole body | Measurements will be obtained at pre-intervention, (0 weeks), mid intervention (14 weeks) and post intervention (40 weeks)
  Whole body T-score. An arbitrary measure, describing the bone mineral density of the subjects relative to a reference value from 30 year old healthy persons.
Change in areal bone mineral density of the lumbar spine (L1-L4) | Measurement will be obtained at pre-intervention, (0 weeks), mid intervention (14 weeks) and post intervention (40 weeks)
  Areal bone mineral density in grams per square centimeter (g/cm2) of the lumbar spine (L1-L4)
Change in T-scores of the lumbar spine (L1-L4) | Measurement will be obtained at pre-intervention, (0 weeks), mid intervention (14 weeks) and post intervention (40 weeks)
  Lumbar spine (L1-L4) T-score. An arbitrary measure, describing the bone mineral density of the subjects relative to a reference value from 30 year old healthy persons.
Change in areal bone mineral density of the bilateral femur regions | Measurement will be obtained at pre-intervention, (0 weeks), mid intervention (14 weeks) and post intervention (40 weeks)
  Areal bone mineral density grams per square centimeter (g/cm2) of the bilateral femur regions
Change in T-scores of the bilateral femur regions | Measurement will be obtained at pre-intervention, (0 weeks), mid intervention (14 weeks) and post intervention (40 weeks)
  T-scores of the bilateral femur regions. An arbitrary measure, describing the bone mineral density of the subjects relative to a reference value from 30 year old healthy persons.
Change in plasma bone turn-over marker (CTX) | Measurement will be obtained at pre-intervention, (0 weeks), mid intervention (14 weeks) and post intervention (40 weeks)
  Carboxy-terminal collagen crosslinks (CTX), measured as μg/L
Change in Plasma bone turn-over marker (P1NP) | Measurement will be obtained at pre-intervention, (0 weeks), mid intervention (14 weeks) and post intervention (40 weeks)
  Procollagen type 1 N-terminal propeptide (P1NP), measured as μg/L
Plasma bone turn-over marker (Osteocalcin) | Measurement will be obtained at pre-intervention, (0 weeks), mid intervention (14 weeks) and post intervention (40 weeks)
  Osteocalcin, measured as μg/L

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nutrition, Exercise and Health, University of Copenhagen, Copenhagen, Capital Region of Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://nexs.ku.dk/forskning/bevaegelse-neurovidenskab/projekter/bevaegelse-samvaer-og-livsduelighed/